CLINICAL TRIAL: NCT05350748
Title: Comprehensive Molecular and Clinical Evaluation of Pediatric and Adult MDS
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000661; 000661-C
Record Dates: First submitted 2022-04-21; First posted 2022-04-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01-14

CONDITIONS: Myelodysplastic Syndromes
Keywords: Heterogenous Stem Cell Disorders; Gene Mutations; Dysplasia; cytopenias; Malignancies; Acute Myeloid Leukemia; Natural History
MeSH Terms: conditions — Myelodysplastic Syndromes; Cytopenia; Neoplasms; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants with myelodysplastic syndromes and associated malignancies
- Cohort 2: Participants (controls) without MDS or associated malignancies, contributing bone marrow

SUMMARY:
Background:

Myelodysplastic syndromes (MDS) occur when the cells that make blood cells are abnormal. There are limited treatment options for MDS. Researchers want to learn more through this natural history study so they can develop better treatments.

Objective:

To study the natural course of MDS and MDS/myeloproliferative neoplasms (MPN) and collect biological samples that can help researchers understand the disease.

Eligibility:

People with suspected or confirmed MDS or MDS/MPN. Healthy donors are also needed. They can be people who are scheduled to donate bone marrow at NIH for a relative, or they may be providing bone marrow in another study.

Design:

Participants will be screened with a medical history.

Participants will have a physical exam. They will give blood and urine samples. They will discuss their symptoms, medications, and ability to perform their normal activities. They will complete surveys about how they are feeling.

Participants will have a bone marrow biopsy. A needle will be inserted through a small cut. Bone marrow will be removed. A small piece of bone may be removed.

Participants may have an optional skin biopsy.

Participants may give optional saliva and stool samples. They may collect these samples at home and mail them to NIH.

Participants may undergo optional apheresis. One or two needles or intravenous (IV) lines will be placed in their arm, neck, or groin veins. Blood will be removed. A machine will separate out the white cells. The rest of the blood will be returned to the participant.

Participants will be contacted for follow-up once a year for up to 20 years.

Healthy donors will have marrow collected for this study during their scheduled procedure with no follow-up.

DETAILED DESCRIPTION:
Background:

* Myelodysplastic syndromes (MDS) are heterogenous stem cell disorders characterized by ineffective hematopoiesis resulting in cellular dysplasia, peripheral cytopenias, and increased risk for transformation to acute myeloid leukemia (AML).
* There are limited treatments options, all of which have unimpressive response rates and limited response durations, with the only potential cure being hematopoietic stem cell transplant (HSCT). Unfortunately, as a disease of the elderly (average age of diagnosis >65 years), most participants are not eligible for HSCT due to advanced age and other comorbidities.
* It is critical we further elucidate the processes that lead to disease manifestation in an effort to develop novel therapeutic strategies and to alter the natural history of the disease.
* Chronic inflammation is central to disease pathology, as evidenced by pro-inflammatory cytokines in the bone marrow milieu, transcriptional upregulation of inflammatory genes, and dysregulation of innate immune signaling pathways.
* We hypothesize the chronic inflammation drives MDS pathogenesis and may be exploited therapeutically. Further, we anticipate the correlatives proposed here to be used not only to uncover critical disease driving pathways, but also to potentially reveal disease and treatment response biomarkers, as well to better refine both diagnosis and prognosis.

Objectives:

- To characterize the natural history of myelodysplastic syndromes (MDS) and to assess overall and progression free survival

Eligibility:

Participants with MDS

* Either sex, any age
* Histologically or cytologically suspected or confirmed MDS, MDS/MPN, (MDS/MPN- RS-T, MDS/MPN-U, CMML, aCML) or sAML with antecedent MDS or MDS/MPN

OR

* diagnosis with a precursor condition that is associated with a risk of progression to MDS.
* Any amount of prior therapy and may be currently receiving MDS-directed therapy.
* Must have an identified primary oncologist, hematologist or generalist outside NIH who agrees to manage care and any diagnostic findings provided by this study.

Controls

* Either sex and must be eligible for marrow donation per clinical center requirements.
* No history of hematological malignancies listed as inclusion criteria for the group of participants with MDS or current autoimmune disease
* Control marrow volunteers must be scheduled for bone marrow harvest for clinical application, or if evaluated for malignancy, have a bone marrow aspirate scheduled to rule out bone marrow involvement at which time additional samples will be taken as controls for the research purposes of this study.

Design:

* This is a natural history and biospecimen acquisition protocol for participants with Myelodysplastic Syndromes (MDS).
* In addition, we will perform a comprehensive research analysis based on the hypothesis that chronic inflammation in MDS arising from a variety of contributors results in hematopoietic differentiation and maturation blocks leading to dysplasia, cytopenias, and disease progression, and that these may be exploited for novel therapeutic targeting strategies.
* This is a single site (Clinical Center) study that will accrue 1000 MDS participants and 100 marrow controls (transplant donor or non-involved malignancy) volunteers over a 20-year study accrual duration.
* Diagnostic testing will be performed as is routine for these participants in addition to planned research correlative analyses. Follow-up will occur approximately annually to assess status and survival.

ELIGIBILITY:
* INCLUSION CRITERIA - MDS Participants
* Either sex, any age.
* Histologically or cytologically suspected or confirmed myelodysplastic syndromes (MDS), myelodysplastic syndromes/myeloproliferative neoplasms (MDS/MPN), MDS/myeloproliferative neoplasm with ringed sideroblasts and thrombocytosis (MDS/MPN-RS-T), myelodysplastic syndromes/myeloproliferative neoplasms unclassified (MDS/MPN-U), chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), secondary acute myeloid leukemia (sAML) with antecedent MDS or MDS/MPN, or participants who have precursor conditions that are associated with a risk of progression to MDS, including but not limited to clonal hematopoiesis of indeterminate potential (CHIP) and clonal cytopenia of unknown significance (CCUS).
* Participants may have had any amount of prior therapy and may be receiving MDS-directed therapy at time of enrollment.
* Participants must have an identified primary oncologist, hematologist or generalist outside of NIH who agrees to manage participant care and any diagnostic findings provided by this study.

INCLUSION CRITERIA - Marrow Control Donor Participants

* Either sex, and must be eligible for marrow donation per NIH Clinical Center requirements.
* No history of hematological malignancies as listed as inclusion in 'Inclusion Criteria - MDS Participants' or current autoimmune disease.
* Must be scheduled for bone marrow harvest for clinical application (e.g., marrow donation); or, if being evaluated for malignancy, have a clinical bone marrow aspirate scheduled (e.g., to rule out bone marrow involvement).

INCLUSION CRITERIA - All Participants

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability of participant or parent/guardian to understand and the willingness to sign a written consent document.

EXCLUSION CRITERIA - All Participants

-Uncontrolled intercurrent illness, psychiatric illness, or other that would limit compliance with study requirements, or at the investigator s discretion.

Ages: 1 Day to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Either sex, any age for participants with MDS. Either sex, aged at least 1 month and >=12kg for bone marrow controls.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2041-09-20 (Estimated); Study Completion 2042-05-01 (Estimated)

PRIMARY OUTCOMES:
characterize the natural history of myelodysplastic syndromes (MDS) and to assess overall and progression free survival | 5 years
  report the overall survival and progression status of participants

SECONDARY OUTCOMES:
acquire biospecimens from MDS patients and controls to perform comprehensive research analyses | Ongoing throughout study
  report the number of participants that have provided at least one of the biospecimens described in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Kathy L McGraw, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI.@@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000661-C.html